CLINICAL TRIAL: NCT03700320
Title: A Phase 3, Multicenter, Randomized, Open-label Study to Evaluate the Long-term Safety and Tolerability of Oral Atogepant for the Prevention of Migraine in Participants With Episodic Migraine
Brief Title: Study to Evaluate the Safety and Tolerability of Treatment With Atogepant 60 mg Daily for the Prevention of Migraine in Participants With Episodic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3101-302-002
Record Dates: First submitted 2018-09-25; First posted 2018-10-09 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Episodic Migraine
MeSH Terms: interventions — Standard of Care; atogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral SOC Migraine Preventive Medication (Active Comparator): Oral standard of care (SOC) medication recognized as safe and effective for the prevention of migraine, based on investigator's judgement in consultation with the participant.
  Interventions: Drug: Standard of Care (SOC) Migraine Preventive Medication
- Atogepant 60 mg (Experimental): Atogepant 60 mg tablet taken orally, once daily for 52 weeks.
  Interventions: Drug: Atogepant

INTERVENTIONS:
Drug: Standard of Care (SOC) Migraine Preventive Medication — Standard of care medication selected based on investigator's judgement, recognized as safe and effective for the prevention of migraine.
  Arms: Oral SOC Migraine Preventive Medication
Drug: Atogepant — Atogepant tablets taken orally, once daily for 52 weeks.
  Arms: Atogepant 60 mg

SUMMARY:
This study will evaluate safety and tolerability of treatment with atogepant for the prevention of episodic migraine over the course of one year.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and participant privacy information (e.g., written authorization for use and release of health and research study information) obtained from the participant prior to initiation of any study-specific procedures.
* Participant is a candidate to be prescribed at least one of the protocol-defined acceptable oral SOC migraine prevention medications and the participant is willing to accept SOC treatment.
* Participants must be using a medically acceptable and effective method of birth control during the course of the entire study,
* At least a 1-year history of migraine with or without aura consistent with a diagnosis
* Age of the participant at the time of migraine onset < 50 years
* History of 4 to 14 migraine days per month on average in the 3 months prior to Visit 1

Exclusion Criteria:

* Difficulty distinguishing migraine headaches from tension-type or other headaches
* Has a history of migraine accompanied by diplopia or decreased level of consciousness or retinal migraine
* Has a current diagnosis of chronic migraine (CM), new persistent daily headache, trigeminal autonomic cephalgia (e.g., cluster headache), or painful cranial neuropathy
* ≥ 15 headache days per month on average across the 3 months prior to Visit 1
* Usage of opioids or barbiturates > 2 days/month, triptans or ergots ≥ 10 days/month, or simple analgesics (e.g., aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen) ≥ 15 days/month in the 3 months prior to Visit 1 per investigator's judgment, or during the baseline period. For all participants, barbiturates are excluded 30 days prior to screening and during the baseline period. For participants randomized to atogepant, barbiturates are excluded through the duration of the study as well
* Female participant is pregnant, planning to become pregnant during the course of the study, or currently lactating. Women of childbearing potential must have a negative urine pregnancy test
* Any clinically significant hematologic, endocrine, pulmonary, renal, hepatic, gastrointestinal (GI), or neurologic disease
* Hypertension as defined by sitting systolic blood pressure (BP) > 160 millimeter of mercury (mm Hg) or sitting diastolic BP > 100 mm Hg at Visits 1 or Visit 2. Vital sign measurements that exceed these limits may be repeated only once.
* At Visit 1, a user of recreational or illicit drugs or has had a history within the past year of drug or alcohol abuse or dependence
* History of any GI prior procedures or GI conditions (e.g., diarrhea syndromes, inflammatory bowel disease) that may affect the absorption or metabolism of atogepant; participants with prior gastric bariatric interventions (e.g., Lap Band) which have been reversed are not excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Trugman, MD, Study Director — Allergan
Locations (112):
- United States (112):
  - Clinical Research Advantage, Inc./Simon Williamson Clinic, PC, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Synexus Clinical Research US, Inc./East Valley Family Physicians PLC, Chandler, Arizona
  - Synexus Clinical Research US, Inc./Desert Clinical Research, LLC, Mesa, Arizona
  - Synexus Clinical Research US, Inc./Central Phoenix Medical Clinic, LLC, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Hope Clinical Research, Canoga Park, California
  - Pharmacology Research Institute, Encino, California
  - Sun Valley Research Center, Inc., Imperial, California
  - Irvine Center for Clinical Research, Irvine, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - Synergy San Diego, Lemon Grove, California
  - Collaborative Neuroscience Network, LLC., Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pacific Research Partners, LLC, Oakland, California
  - Excell Research, Inc., Oceanside, California
  - Desert Valley Research, Redlands, California
  - Medical Center for Clinical Research, San Diego, California
  - California Research Foundation, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Encompass Clinical Research, Spring Valley, California
  - Synexus Clinical Research US, Inc., Vista, California
  - Diablo Clinical Research, Inc, Walnut Creek, California
  - Delta Waves, Inc., Colorado Springs, Colorado
  - Advanced Neurosciences Research, LLC, Fort Collins, Colorado
  - MD Clinical, Hallandale, Florida
  - Infinity Clinical Research, Hollywood, Florida
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Meridien Research, Maitland, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Bioclinica Research, Orlando, Florida
  - Infinity Clinical Research LLC, Sunrise, Florida
  - Meridien Research, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Synexus Clinical Research US, Inc., Atlanta, Georgia
  - Atlanta Center for Clinical Research, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - MidAmerica Neuroscience Research Foundation dba Rowe Neurology Institute, Lenexa, Kansas
  - Kansas Institute of Research, Overland Park, Kansas
  - Phoenix Medical Research, Inc., Prairie Village, Kansas
  - Kentucky Pediatric Research, Bardstown, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Community Clinical Research Network, Marlborough, Massachusetts
  - Michigan Headache & Neurological Institute, Ann Arbor, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - ClinVest, Springfield, Missouri
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Synexus Clinical Research US, Inc, Omaha, Nebraska
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institutes, Berlin, New Jersey
  - Amici Clinical Research, Raritan, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Dent Neurosciences Research Center, Amherst, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Synexus Clinical Research US, Inc., Jamaica, New York
  - Central New York Clinical Research, Manlius, New York
  - Rochester Clinical Research, Rochester, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Plains Clinical Medical Clinic, LLC, Fargo, North Dakota
  - Synexus Clinical Research US, Inc., Akron, Ohio
  - Synexus Clinical Research US, Inc., Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Ohio Clinical Research, LLC, Willoughby Hills, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Radiant Research, Inc., Anderson, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Meridian Clinical Research, LLC, Dakota Dunes, South Dakota
  - Volunteer Research Group, Knoxville, Tennessee
  - CNS Healthcare - Memphis, Memphis, Tennessee
  - Trinity Clinical Research, Tullahoma, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Tekton Research, Inc, Austin, Texas
  - DiscoveResearch, Inc., Bryan, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Earle Research, Houston, Texas
  - Research Trials WorldWide, LLC, Humble, Texas
  - Synexus Clinical Research US, Inc., San Antonio, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - J. Lewis Research, Inc./Foothill Family Clinic Draper, Draper, Utah
  - Advanced Research Institute, Ogden, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Women's: Health, Research, Seattle, Washington
  - SSM Dean Health Research, Madison, Wisconsin

REFERENCES:
- [Derived] Peterlin BL, Bond DS, Ailani J, Dodick DW, Liu Y, De Abreu Ferreira R, Smith JH, Dabruzzo B, Goadsby PJ, Trugman JM. Weight loss with atogepant during the preventive treatment of migraine: A pooled analysis. Cephalalgia. 2024 Dec;44(12):3331024241299753. doi: 10.1177/03331024241299753. PMID 39648629
- [Derived] Lipton RB, Nahas SJ, Pozo-Rosich P, Bilchik T, McAllister P, Finnegan M, Liu Y, Chalermpalanupap N, Dabruzzo B, Dodick DW. Sustained response to atogepant in episodic migraine: post hoc analyses of a 12-week randomized trial and a 52-week long-term safety trial. J Headache Pain. 2024 May 21;25(1):83. doi: 10.1186/s10194-024-01783-6. PMID 38773375
- [Derived] Rizzoli P, Marmura MJ, Robblee J, McVige J, Sacco S, Nahas SJ, Ailani J, De Abreu Ferreira R, Ma J, Smith JH, Dabruzzo B, Ashina M. Safety and tolerability of atogepant for the preventive treatment of migraine: a post hoc analysis of pooled data from four clinical trials. J Headache Pain. 2024 Mar 11;25(1):35. doi: 10.1186/s10194-024-01736-z. PMID 38462625
- [Derived] Lipton RB, Halker Singh RB, Mechtler L, McVige J, Ma J, Yu SY, Stokes J, Dabruzzo B, Gandhi P, Ashina M. Patient-reported migraine-specific quality of life, activity impairment and headache impact with once-daily atogepant for preventive treatment of migraine in a randomized, 52-week trial. Cephalalgia. 2023 Aug;51(8):3331024231190296. doi: 10.1177/03331024231190296. PMID 37638400
- [Derived] Boinpally R, McNamee B, Yao L, Butler M, McGeeney D, Borbridge L, Periclou A. A Single Supratherapeutic Dose of Atogepant Does Not Affect Cardiac Repolarization in Healthy Adults: Results From a Randomized, Single-Dose, Phase 1 Crossover Trial. Clin Pharmacol Drug Dev. 2021 Sep;10(9):1099-1107. doi: 10.1002/cpdd.940. Epub 2021 May 4. PMID 33942560
- [Derived] Min KC, Kraft WK, Bondiskey P, Colon-Gonzalez F, Liu W, Xu J, Panebianco D, Mixson L, Dockendorf MF, Matthews CZ, Boinpally R. Atogepant Is Not Associated With Clinically Meaningful Alanine Aminotransferase Elevations in Healthy Adults. Clin Transl Sci. 2021 Mar;14(2):599-605. doi: 10.1111/cts.12917. Epub 2020 Nov 24. PMID 33142014

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral SOC Migraine Preventive Medication | Atogepant 60 mg
Started | 198 | 546
Safety Population; Received Treatment | 196 | 543
Entered Safety Follow-up | 159 | 472
Completed | 136 | 373
Not Completed | 62 | 173
Not completed — Adverse Event | 5 | 31
Not completed — Lack of Efficacy | 2 | 5
Not completed — Withdrawal by Subject | 29 | 75
Not completed — Lost to Follow-up | 16 | 23
Not completed — Pregnancy | 2 | 4
Not completed — Protocol Deviation | 7 | 31
Not completed — Non-compliance with Study Drug | 1 | 3
Not completed — Reason not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received ≥1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral SOC Migraine Preventive Medication | Atogepant 60 mg | Total
Number analyzed (Participants) | 196 | 543 | 739
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (12.09) | 42.5 (12.03) | 42.2 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 479 | 651
  Male | 24 | 64 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 83 | 112
  Not Hispanic or Latino | 166 | 460 | 626
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 5 | 12 | 17
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 38 | 100 | 138
  White | 145 | 416 | 561
  More than one race | 5 | 10 | 15
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is an AE that occurs or worsens after receiving investigational study drug.
Time Frame: From first dose up to the end of study (median treatment of 52 weeks) + 4 weeks follow-up
Population: Safety Population included all participants who received ≥1 dose of study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Oral SOC Migraine Preventive Medication | Atogepant 60 mg
Number analyzed (Participants) | 196 | 543
percentage of participants | 78.6 | 67.0

2. Secondary Outcome: Percentage of Participants With Clinically Significant Laboratory Values as Assessed by the Investigator
Description: Laboratory tests included tests of hematology, chemistry, and urinalysis. The investigator determined if the results were potentially clinically significant (PCS). Only categories with at least one participant are reported.
Time Frame: From first dose up to the end of study (median treatment of 52 weeks) + 4 weeks follow-up
Population: Safety Population included all participants who received ≥1 dose of study intervention. Number analyzed is the number of participants with non-missing non-PCS baseline value and ≥1 post-baseline parameter assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Oral SOC Migraine Preventive Medication | Atogepant 60 mg
Number analyzed (Participants) | 196 | 543
percentage of participants
  Eosinophils Absolute Cell Count (10^9/liter (L)): >2.0 × upper limit of normal (ULN): number analyzed (Participants) | 190 | 531
  Eosinophils Absolute Cell Count (10^9/liter (L)): >2.0 × upper limit of normal (ULN) | 0.0 | 0.6
  Hematocrit (RATIO): <0.9 × lower limit of normal (LLN): number analyzed (Participants) | 190 | 531
  Hematocrit (RATIO): <0.9 × lower limit of normal (LLN) | 1.6 | 1.7
  Hematocrit (RATIO): >1.1 × ULN: number analyzed (Participants) | 190 | 531
  Hematocrit (RATIO): >1.1 × ULN | 0.0 | 0.2
  Hemoglobin (gram (g)/L): <0.9 × LLN: number analyzed (Participants) | 184 | 521
  Hemoglobin (gram (g)/L): <0.9 × LLN | 3.3 | 3.1
  Lymphocytes Absolute Cell Count (10^9/L): <0.7 × LLN: number analyzed (Participants) | 189 | 530
  Lymphocytes Absolute Cell Count (10^9/L): <0.7 × LLN | 0.5 | 0.8
  Lymphocytes Absolute Cell Count (10^9/L): >1.3 × ULN: number analyzed (Participants) | 189 | 530
  Lymphocytes Absolute Cell Count (10^9/L): >1.3 × ULN | 0.5 | 0.2
  Monocytes Absolute Cell Count (10^9/L): <0.5 × LLN: number analyzed (Participants) | 190 | 531
  Monocytes Absolute Cell Count (10^9/L): <0.5 × LLN | 1.1 | 0.2
  Neutrophils Absolute Cell Count (10^9/L): <0.7 × LLN: number analyzed (Participants) | 189 | 523
  Neutrophils Absolute Cell Count (10^9/L): <0.7 × LLN | 2.1 | 2.3
  Neutrophils Absolute Cell Count (10^9/L): >1.3 × ULN: number analyzed (Participants) | 189 | 523
  Neutrophils Absolute Cell Count (10^9/L): >1.3 × ULN | 4.8 | 7.1
  Platelet Count (Thrombocytes) (10^9/L): >1.5 × ULN: number analyzed (Participants) | 189 | 531
  Platelet Count (Thrombocytes) (10^9/L): >1.5 × ULN | 0.5 | 0.2
  Red Blood Cell Count (10^12/L): <0.9 × LLN: number analyzed (Participants) | 188 | 529
  Red Blood Cell Count (10^12/L): <0.9 × LLN | 3.2 | 2.1
  White Blood Cell Count (10^9/L): <0.9 × LLN: number analyzed (Participants) | 187 | 526
  White Blood Cell Count (10^9/L): <0.9 × LLN | 3.2 | 4.6
  White Blood Cell Count (10^9/L): >1.5 × ULN: number analyzed (Participants) | 187 | 526
  White Blood Cell Count (10^9/L): >1.5 × ULN | 1.1 | 0.6
  Alanine Aminotransferase (serum glutamic-pyruvic transaminase (SGPT)) (Unit (U)/L): ≥3.0 × ULN: number analyzed (Participants) | 190 | 530
  Alanine Aminotransferase (serum glutamic-pyruvic transaminase (SGPT)) (Unit (U)/L): ≥3.0 × ULN | 1.6 | 1.9
  Aspartate Aminotransferase (serum glutamic-oxaloacetic transaminase (SGOT)) (U/L): ≥3.0 × ULN: number analyzed (Participants) | 190 | 529
  Aspartate Aminotransferase (serum glutamic-oxaloacetic transaminase (SGOT)) (U/L): ≥3.0 × ULN | 2.1 | 1.5
  Bicarbonate (HCO3) (millimole (mmol)/L): <0.9 × LLN: number analyzed (Participants) | 190 | 531
  Bicarbonate (HCO3) (millimole (mmol)/L): <0.9 × LLN | 1.6 | 0.8
  Bilirubin, Total (micromole (umol)/L): ≥1.5 × ULN: number analyzed (Participants) | 190 | 530
  Bilirubin, Total (micromole (umol)/L): ≥1.5 × ULN | 0.0 | 0.8
  Blood Urea Nitrogen (mmol/L): >1.5 × ULN: number analyzed (Participants) | 190 | 531
  Blood Urea Nitrogen (mmol/L): >1.5 × ULN | 0.5 | 0.4
  Creatine Kinase (U/L): >2.0 × ULN: number analyzed (Participants) | 185 | 525
  Creatine Kinase (U/L): >2.0 × ULN | 14.1 | 9.1
  Creatinine (umol/L): >1.5 × ULN: number analyzed (Participants) | 190 | 531
  Creatinine (umol/L): >1.5 × ULN | 1.1 | 0.4
  Glomerular Filtration Rate(GFR) Estimated Calculation:<60 milliliter(mL)/minute(min)/1.73 meter(m)^2: number analyzed (Participants) | 184 | 503
  Glomerular Filtration Rate(GFR) Estimated Calculation:<60 milliliter(mL)/minute(min)/1.73 meter(m)^2 | 15.2 | 15.9
  Glucose, Non-fasting (mmol/L): <0.8 × LLN: number analyzed (Participants) | 188 | 527
  Glucose, Non-fasting (mmol/L): <0.8 × LLN | 5.3 | 4.2
  Glucose, Non-fasting (mmol/L): >2.0 × ULN: number analyzed (Participants) | 188 | 527
  Glucose, Non-fasting (mmol/L): >2.0 × ULN | 2.1 | 0.8
  Lactate Dehydrogenase (U/L): >3.0 × ULN: number analyzed (Participants) | 189 | 529
  Lactate Dehydrogenase (U/L): >3.0 × ULN | 0.0 | 0.4
  Phosphorus (mmol/L): <0.9 × LLN: number analyzed (Participants) | 190 | 530
  Phosphorus (mmol/L): <0.9 × LLN | 2.1 | 2.6
  Phosphorus (mmol/L): >1.1 × ULN: number analyzed (Participants) | 190 | 530
  Phosphorus (mmol/L): >1.1 × ULN | 0.0 | 0.2
  Potassium (mmol/L): <0.9 × LLN: number analyzed (Participants) | 188 | 525
  Potassium (mmol/L): <0.9 × LLN | 1.1 | 0.8
  Potassium (mmol/L): >1.1 × ULN: number analyzed (Participants) | 188 | 525
  Potassium (mmol/L): >1.1 × ULN | 4.3 | 5.1
  Protein, Total (g/L): <0.9 × LLN: number analyzed (Participants) | 190 | 531
  Protein, Total (g/L): <0.9 × LLN | 3.2 | 1.5
  Uric Acid (Urate) (umol/L): >1.2 × ULN: number analyzed (Participants) | 190 | 531
  Uric Acid (Urate) (umol/L): >1.2 × ULN | 1.6 | 1.1
  Urine Glucose At Least 1+: number analyzed (Participants) | 185 | 526
  Urine Glucose At Least 1+ | 4.3 | 3.0
  Urine Protein: At Least 1+: number analyzed (Participants) | 183 | 497
  Urine Protein: At Least 1+ | 26.2 | 27.4

3. Secondary Outcome: Percentage of Participants With Clinically Significant Electrocardiogram (ECG) Findings as Assessed by the Investigator
Description: A standard 12-lead ECG was performed. The investigator determined if the result was potentially clinically significant. Only categories with at least one participant are reported.
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Oral SOC Migraine Preventive Medication | Atogepant 60 mg
Number analyzed (Participants) | 196 | 543
percentage of participants
  PR Interval, Single Beat millisecond (msec): ≥250: number analyzed (Participants) | 179 | 513
  PR Interval, Single Beat millisecond (msec): ≥250 | 0.0 | 0.2
  QTcB Interval, Single Beat (msec): Increase >60 from Baseline (BL): number analyzed (Participants) | 180 | 514
  QTcB Interval, Single Beat (msec): Increase >60 from Baseline (BL) | 0.6 | 0.4
  QTcF Interval, Single Beat (msec): Increase >60 from BL: number analyzed (Participants) | 180 | 514
  QTcF Interval, Single Beat (msec): Increase >60 from BL | 0.6 | 0.0

4. Secondary Outcome: Percentage of Participants With Clinically Significant Vital Sign Measurements as Assessed by the Investigator
Description: Vital sign measurements included sitting and standing blood pressure (BP), sitting and standing pulse rate, respiratory rate, temperature, and body weight. The investigator determined if the results were clinically significant. Only categories with at least one participant are reported.
Time Frame: From first dose up to the end of study (median treatment of 52 weeks + 4 weeks follow-up)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Oral SOC Migraine Preventive Medication | Atogepant 60 mg
Number analyzed (Participants) | 196 | 543
percentage of participants
  Systolic Blood Pressure (SBP) Sitting (millimeter of mercury(mmHg)):≤90 and Decrease of ≥20 from BL: number analyzed (Participants) | 190 | 531
  Systolic Blood Pressure (SBP) Sitting (millimeter of mercury(mmHg)):≤90 and Decrease of ≥20 from BL | 3.7 | 2.6
  SBP Sitting (mmHg): ≥180 and Increase of ≥20 from BL: number analyzed (Participants) | 190 | 531
  SBP Sitting (mmHg): ≥180 and Increase of ≥20 from BL | 0.0 | 0.4
  SBP Standing (mmHg): ≤90 and Decrease of ≥20 from BL: number analyzed (Participants) | 190 | 531
  SBP Standing (mmHg): ≤90 and Decrease of ≥20 from BL | 5.8 | 3.4
  SBP Standing (mmHg): ≥180 and Increase of ≥20 from BL: number analyzed (Participants) | 190 | 531
  SBP Standing (mmHg): ≥180 and Increase of ≥20 from BL | 0.0 | 0.6
  Standing - Sitting SBP (mmHg): ≤-20: number analyzed (Participants) | 189 | 526
  Standing - Sitting SBP (mmHg): ≤-20 | 13.8 | 11.4
  Diastolic Blood Pressure (DBP) Sitting (mmHg): ≤50 and Decrease of ≥15 from BL: number analyzed (Participants) | 190 | 531
  Diastolic Blood Pressure (DBP) Sitting (mmHg): ≤50 and Decrease of ≥15 from BL | 3.2 | 0.6
  DBP Sitting (mmHg): ≥105 and Increase of ≥15 from BL: number analyzed (Participants) | 190 | 531
  DBP Sitting (mmHg): ≥105 and Increase of ≥15 from BL | 1.1 | 2.3
  DBP Standing (mmHg): ≤50 and Decrease of ≥15 from BL: number analyzed (Participants) | 190 | 531
  DBP Standing (mmHg): ≤50 and Decrease of ≥15 from BL | 1.1 | 0.9
  DBP Standing (mmHg): ≥105 and Increase of ≥15 from BL: number analyzed (Participants) | 190 | 531
  DBP Standing (mmHg): ≥105 and Increase of ≥15 from BL | 5.8 | 4.0
  Standing - Sitting DBP (mmHg): ≤-15: number analyzed (Participants) | 189 | 528
  Standing - Sitting DBP (mmHg): ≤-15 | 10.1 | 8.7
  Pulse Rate (PR) Sitting (beats/min): ≤50 and Decrease of ≥15 from BL: number analyzed (Participants) | 190 | 531
  Pulse Rate (PR) Sitting (beats/min): ≤50 and Decrease of ≥15 from BL | 1.6 | 1.1
  PR Standing (beats/min): ≤50 and Decrease of ≥15 from BL: number analyzed (Participants) | 190 | 531
  PR Standing (beats/min): ≤50 and Decrease of ≥15 from BL | 0.0 | 0.2
  PR Standing (beats/min): ≥120 and Increase of ≥15 from BL: number analyzed (Participants) | 190 | 531
  PR Standing (beats/min): ≥120 and Increase of ≥15 from BL | 2.6 | 1.3
  Standing - Sitting PR (beats/min): ≥25: number analyzed (Participants) | 190 | 528
  Standing - Sitting PR (beats/min): ≥25 | 6.3 | 10.0
  Weight (kg): Decrease of ≥7% from BL: number analyzed (Participants) | 190 | 531
  Weight (kg): Decrease of ≥7% from BL | 14.7 | 24.1
  Weight (kg): Increase of ≥7% from BL: number analyzed (Participants) | 190 | 531
  Weight (kg): Increase of ≥7% from BL | 12.6 | 7.3

5. Secondary Outcome: Number of Participants With Most Severe Columbia-Suicide Severity Rating Scale (C-SSRS) Assessing Suicidal Ideation or Suicidal Behavior
Description: The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior. Suicidal ideation was classified on a 5-item scale: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent). Suicidal behavior is classified on a 5-item scale: 0 (no suicidal behavior), 1 (preparatory acts or behavior), 2 (aborted attempt), 3 (interrupted attempt), and 4 (actual attempt). More than 1 classification can be selected provided they represent separate episodes. (Minimum total score 0, maximum total score 5; higher total scores indicate more suicidal ideation and/or suicidal behavior). Only the most severe suicidal ideation and the most severe suicidal behavior counted during the treatment period for at least 1 participant are reported.
Time Frame: Up to Week 52
Population: Safety Population included all participants who received ≥1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral SOC Migraine Preventive Medication | Atogepant 60 mg
Number analyzed (Participants) | 196 | 543
Participants
  Suicidal Ideation (SI): Wish to be Dead | 4 | 0
  SI: Non-Specific Active Suicidal Thoughts | 1 | 2
  SI: Active SI with Some Intent to Act, Without Specific Plan | 0 | 1
  SI: Active SI With Specific Plan and Intent | 0 | 2
  Suicidal Behavior (SB): Actual Attempt | 0 | 2

ADVERSE EVENTS:
Time Frame: From first dose up to the end of study (median treatment of 52 weeks + 4 weeks follow-up)
Description: All-cause Mortality: Intent-to-treat (ITT) Population included all randomized participants. Adverse Events: Safety Population included all participants who received ≥1 dose of study intervention.
Arm/Group | Oral SOC Migraine Preventive Medication | Atogepant 60 mg
All-Cause Mortality (participants affected / at risk) | 0/198 | 2/546
Serious Adverse Events (participants affected / at risk) | 7/196 | 24/543
Other Adverse Events (participants affected / at risk) | 91/196 | 197/543
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Oral SOC Migraine Preventive Medication (N=196) | Atogepant 60 mg (N=543)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/172 | 1/479 — Number of participants at risk are female participants as this adverse event is specific to females.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Status migrainosus (Nervous system disorders) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1
Device malfunction (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0/172 | 1/479 — Number of participants at risk are female participants as this adverse event is specific to females.
Uterine haemorrhage (Reproductive system and breast disorders) | 0/172 | 1/479 — Number of participants at risk are female participants as this adverse event is specific to females.
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Victim of crime (Social circumstances) | 0 | 1
Victim of homicide (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral SOC Migraine Preventive Medication (N=196) | Atogepant 60 mg (N=543)
Constipation (Gastrointestinal disorders) | 6 | 39
Nausea (Gastrointestinal disorders) | 12 | 34
Fatigue (General disorders) | 12 | 14
Upper respiratory tract infection (Infections and infestations) | 24 | 56
Urinary tract infection (Infections and infestations) | 9 | 28
Nasopharyngitis (Infections and infestations) | 10 | 24
Weight increased (Investigations) | 11 | 7
Dizziness (Nervous system disorders) | 22 | 17
Paraesthesia (Nervous system disorders) | 12 | 8
Anxiety (Psychiatric disorders) | 11 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT03700320/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT03700320/SAP_001.pdf